CLINICAL TRIAL: NCT06464666
Title: Association Between Renal Resistive Index(RRI) and AKI(Acute Kidney Injury) in Cardiac Surgery Patients With Cardiopulmonary Bypass (CPB)
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-0439
Record Dates: First submitted 2024-06-10; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Acute Kidney Injury; Renal Resistive Index
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RRI positive group: RRI value higher than 0.7 measured by renal interlobar artery US
  Interventions: Procedure: Renal interlobar artery US
- RRI negative group: RRI value lower than 0.7 measured by renal interlobar artery US
  Interventions: Procedure: Renal inter-lobular artery US

INTERVENTIONS:
Procedure: Renal interlobar artery US — By using convex US transducer, first find interlobar artery. Then get a pulsed wave doppler at renal interlobar artery for similar 3 to 5 waveforms. Measure peak systolic and minimum diastolic velocity and calculate RRI value.
  Groups: RRI positive group
Procedure: Renal inter-lobular artery US — By using convex US transducer, first find interlobar artery. Then get a pulsed wave doppler at renal interlobar artery for similar 3 to 5 waveforms. Measure peak systolic and minimum diastolic velocity and calculate RRI value.
  Groups: RRI negative group

SUMMARY:
AKI(Acute Kidney Injury) is a common complication after cardiac surgery which is associated with increased mortality and morbidity. The conventiional marker for detecting AKI is serum creatinine, however, which has many limits. RRI(Renal Resistive Index) is a non-invasive test measured by ultrasound and could be a useful tool to evaulate renal insult in the early phase. Early detection of renal insult and prevention of progression to AKI can contribute to reduing mortality and morbidity in cardiac surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years and older scheduled for cardiac surgery using CPB

Exclusion Criteria:

* Emergency opeartion, pre-operative shock status requiring vasopressor or inotropics, s/p kidney transplant patients, CKD stage 4 and 5 patients, patients who have renal artery stenosis or history of renal artery stent implantation, patients who have ascites with Child-Pugh classification B or C, In case of CPB weaning failure, In case of poor lung function and PaO2 or PaCO2 cannot be maintained within normal range.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Association between renal resistive index(RRI) and AKI(Acute Kidney Injury) in cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
post-operative AKI incidence | within first 1 week after surgery
  The definition of AKI refers to Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury Work Group. KDIGO Clinical Practice Guideline for Acute Kidney Injury.

SECONDARY OUTCOMES:
Major adverse kidney outcome (MAKE) 30 | within first 1 month after surgery
  MAKE30 includes new dialysis, eGFR decrease more than 25% from the baseline, and mortality

IPD SHARING:
Plan to Share IPD: No